CLINICAL TRIAL: NCT00005831
Title: Phase II Evaluation of Trastuzumab (Herceptin), Paclitaxel, Carboplatin, and Gemcitabine in the Treatment of Advanced Urothelial Cancer
Brief Title: Trastuzumab and Combination Chemotherapy in Treating Patients With Locally Recurrent or Metastatic Urinary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03187; UMCC-9955; U01CA062487 (NIH); N01CM17101 (NIH); CDR0000067845 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Bladder Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Squamous Cell Carcinoma of the Bladder; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Trastuzumab; Paclitaxel; Taxes; Carboplatin; Gemcitabine

ARMS (1):
- Treatment (trastuzumab, combination chemotherapy) (Experimental): Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15; paclitaxel IV over 3 hours and carboplatin IV over 15 minutes on day 1; and gemcitabine IV over 30 minutes on days 1 and 8. Courses repeat every 3 weeks. Patients achieving a complete response (CR) receive 3 courses past CR. Patients achieving a partial response or stable disease continue on therapy until CR or disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Drug: paclitaxel; Drug: carboplatin; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining trastuzumab with combination chemotherapy in treating patients who have locally recurrent or metastatic urinary tract cancer. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with combination chemotherapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the toxicity of the combination of Herceptin, paclitaxel, carboplatin, and gemcitabine in patients with metastatic or locally recurrent urothelial cancers who overexpress HER2.

SECONDARY OBJECTIVES:

I. The complete and partial response rates. II. The median and overall survival. III. To prospectively evaluate the percentage of patients with metastatic/recurrent bladder cancer who overexpress HER2 histologically (by immunohistochemistry and FISH) and serologically.

IV. To generate preliminary data on response to other therapy and survival for Her2 negative patients.

OUTLINE:

Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15; paclitaxel IV over 3 hours and carboplatin IV over 15 minutes on day 1; and gemcitabine IV over 30 minutes on days 1 and 8. Courses repeat every 3 weeks. Patients achieving a complete response (CR) receive 3 courses past CR. Patients achieving a partial response or stable disease continue on therapy until CR or disease progression or unacceptable toxicity.

Patients are followed for disease progression and survival. Patients with HER2-negative disease are not eligible for treatment but are followed every 6 months for response and survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of urothelial carcinoma (TCC or Squamous) that is either metastatic or locally recurrent and not curable by surgery or radiation therapy; patients must have HER2 overexpression as documented by ANY of the following: 1. 2+ or 3+ staining by immunohistochemistry, or 2. a positive FISH score defined as > 2 with the Vysis system or > 4 with the Ventana system, or 3. an elevated serum HER2 of > 16 ng/ml using the OSDI assay; please note:

  * Tissue from either the primary or metastatic site must be tested for HER2 status determination
  * All patients must have a blood sample drawn for HER2 serologic testing
  * If the available tissue is from the primary tumor and is HER2 negative and if the serum is negative, to qualify for the study a biopsy of a metastatic site should be done and the patient will be eligible ONLY if this demonstrates HER2 over-expression
  * All sites and measurements of disease must be clearly documented in the pre-study forms
  * All prior local or adjuvant systemic therapy including the type of chemotherapy must be clearly documented in the pre-study form Note: Patients with Her-2 negative tumors are not eligible for treatment on this protocol but their response to other therapy and survival will also be evaluated
* Bidimensionally measurable or evaluable disease not previously radiated
* No prior systemic chemotherapy for metastatic disease; patients may have received adjuvant chemotherapy if completed at least 6 months prior to beginning this protocol treatment; type and number of courses of prior chemotherapy must be clearly documented
* A performance status of 0-2 by Southwest Oncology Group criteria and a life expectancy of greater than 12 weeks
* Serum creatinine =< 2.0 mg%
* Granulocyte count >= 1,500/mm^3
* Platelet >= 100,000/mm^3
* Total bilirubin =< 1.5 mg/dl
* No significant cardiac disease and must have adequate cardiac function (ejection fraction >= 50% or higher than the lower limit of institutional normal) as determined by a MUGA scan or 2-D echocardiogram within 4 weeks from registration, and no evidence of symptomatic coronary artery disease (baseline EKG must show no active ischemia); patients must not have history of congestive heart failure
* If patients have received prior radiation therapy, disease must be present outside of radiated fields and at least 4 weeks must have elapsed since discontinuation of that therapy; the nadirs of RT leukopenia and thrombocytopenia must be surpassed with evidence of hematologic recovery
* No prior malignancy is allowed, except for adequately treated basal cell (or squamous cell) skin cancer, in situ carcinoma of any site or other cancer for which the patient is currently disease free
* Patient may not have unresolved bacterial infection
* Pregnant or lactating women may not participate; this is to avoid potential harm since the effects of study drugs on the fetus or the nursing infant are not known; women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* HIV -positive patients may not participate; this is to avoid additional complications that immune suppression and HIV infection may cause due to the intense nature of the chemotherapy in this trial
* Timing guidelines for pre-study labs (excluding HER2 determination) and measurements;

  * To be completed within 14 days prior to registration; pre-study labs required for determination of eligibility
  * To be completed within 28 days prior to registration: x-rays, scans or physical examination used for tumor
* All patients must be informed of the investigational nature of this study and must sign an informed consent in accordance with institutional and federal guidelines
* All patients must be registered with the UM Cancer Center Clinical Trials Office at 734-647-8174 (Joanne Goodson) prior to instituting therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2000-03; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Cardiac toxicity rate of this combination using MUGA or 2D ECHO | Up to 7 years
Response rate | Up to 7 years
  The response rate of this regimen will be estimated with a standard error no greater than 7.9%.

SECONDARY OUTCOMES:
Time to disease progression | Up to 7 years
  Kaplan-Meier method will be used for the analysis and graphic presentation of this data.
Survival duration | Up to 7 years
  Kaplan-Meier method will be used for the analysis and graphic presentation of this data.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, Principal Investigator — University of Michigan University Hospital
Locations (1):
- University of Michigan University Hospital, Ann Arbor, Michigan, United States